CLINICAL TRIAL: NCT00750334
Title: A Phase I, Open-Label, Dose-Finding and Food Effect Study of Oral Clofarabine in Previously Treated Adult Patients With Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Oral Clofarabine in Adult Patients With Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated to focus on comparable trial, CLOMDS02507
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOMDS01206
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Oral Clofarabine,; relapsed/refractory MDS,; Myelodysplastic
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): clofarabine Dose Escalation
  Interventions: Drug: clofarabine
- Part B (Experimental): Part B is an open-label, replicated cross-over study in which 12 additional patients will be enrolled and treated at the MTD determined in part A to evaluate the effect of food on the PK disposition of oral clofarabine.
  Interventions: Drug: clofarabine

INTERVENTIONS:
Drug: clofarabine — Drug given Daily x 14 days and 7 days of rest for 21 day cycle
  Arms: Part A
Drug: clofarabine — Drug given Daily X 14 days and 7 days of rest for 21 day cycle
  Arms: Part B

SUMMARY:
This study will be used to determine the maximum tolerated dose of oral clofarabine when administered daily for 14 consecutive days repeated every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed, written informed consent.
* Be at least 18 years old.
* Have a pathologically confirmed MDS and score according to the IPSS at study entry. Pathologic confirmation is the responsibility of the investigator.
* Have been treated previously for MDS as follow: a.Patients must have had at least 1, but no more than 2, prior treatment regimens; b.Patients must not have refractory (i.e., disease progression or no evidence of response while on treatment) to more than 1 prior treatment regimen.
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Be able to comply with study procedures and follow-up examinations.
* Have adequate hepatic and renal function.
* Be non-fertile or agree to use birth control during the study through the end of the last treatment visit and at least 90 days after.

Exclusion Criteria:

* Have had a readjustment of dose and/or schedule of erythropoietin, granulocyte colony stimulating factor(G-CSF) or other growth factors within 8 weeks prior to the first dose of oral clofarabine.
* Have had any other chemotherapy or any investigational therapy for MDS within 4 weeks of the first dose of oral clofarabine.
* Have not recovered to ≤ Grade 2 in severity of any drug-related non-hematologic toxicity prior to the first dose of oral clofarabine.
* Have an uncontrolled systemic fungal, bacterial, viral or other infection. Have a history of serious disease involving the heart.
* Have a clinically significant cardiac assessment at screening or a known family history QT prolongation.
* Currently uses a medication known to prolong the QT interval.
* Have had any prior treatment with clofarabine (IV or oral).
* Have had a diagnosis of another malignancy, unless the patient has been disease free for at least 3 years after completing curative intent therapy except for the following: a. Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment or the condition has been completed. b. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Have prior positive test for the human immunodeficiency virus (HIV).
* Have gastrointestinal disease or prior surgery, which may affect the ability of the patient to absorb oral clofarabine.
* Is currently participating in another concurrent investigational protocol that is not restricted to data and/or sample collection for patient demographic and/or disease purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated dose levels | First Cycle

SECONDARY OUTCOMES:
PK profile | After MTD is established
Food effect on profile | After MTD is established
Activity of clofarabine in this dosing regimen | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Malignant Hematology Administration, H. Lee Moffitt Cancer Center, Tampa, Florida
  - Division of Hematology Mayo Clinic, Rochester, Minnesota
  - Cancer Care Centers of South Texas, San Antonio, Texas